CLINICAL TRIAL: NCT03536637
Title: A Study of Tolerability, Safety, And Efficacy, of DMT310 In Patients With Acne Vulgaris
Brief Title: DMT310-001 Topical in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMT310-001
Record Dates: First submitted 2018-05-02; First posted 2018-05-25 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2018-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Study Treatment 1 (Experimental): DMT310 Powder mixed with Hydrogen Peroxide
  Interventions: Drug: DMT310; Drug: Hydrogen Peroxide
- Study Treatment 2 (Experimental): DMT310 Powder mixed with Placebo Diluent
  Interventions: Drug: DMT310
- Study Treatment 3 (Experimental): Placebo powder mixed with Hydrogen Peroxide
  Interventions: Drug: Hydrogen Peroxide; Drug: Placebo
- Control (Placebo Comparator): Placebo powder mixed with Placebo Diluent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMT310 — Topical Powder
  Arms: Study Treatment 1; Study Treatment 2
Drug: Hydrogen Peroxide — Liquid Diluent
  Arms: Study Treatment 1; Study Treatment 3
Drug: Placebo — Placebo Topical Powder
  Arms: Control; Study Treatment 3

SUMMARY:
The objective is to evaluate the tolerability, safety, and efficacy of DMT310 topical powder mixed with diluent in male and female patients with moderate to severe facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or non-pregnant female at least 18 years of age.
* Clinical diagnosis of moderate to severe acne vulgaris as determined by:

Investigator's Global Assessment (IGA) at Randomization Patient has at least 20 but not more than 50 inflammatory lesions on the face Patient has at least 20 but not more than 100 noninflammatory lesions on the face

* Patient is willing to apply the Investigational Product as directed
* Patient is willing and able to comply with the protocol

Exclusion Criteria:

* Patient is pregnant or planning to become pregnant
* Patient is taking a topical therapy on the face which may affect the patient's acne

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by lesion counts | 12 weeks
  Inflammatory and Noninflammatory
Efficacy as measured by Investigator Global Assessment (IGA) | 12 weeks
  0 None No evidence of facial acne vulgaris
  1. Minimal Few noninflammatory lesions (comedones) are present; a few inflammatory lesions(papules/pustules) may be present; no nodulo-cystic lesions are allowed)
  2. Mild Several to many noninflammatory lesions (comedones) are present; a few inflammatory lesions (papules/pustules) are present; no nodulo-cystic lesions are allowed
  3. Moderate Many noninflammatory (comedones) and inflammatory lesions (papules/pustules) are present; no nodulo-cystic lesions are allowed
  4. Severe Significant degree of inflammatory disease; papules/pustules are a predominant feature; a few nodulo-cystic lesions may be present; comedones may be present

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 12 weeks
  Incidence of adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Dermata Investigational Site, San Diego, California
  - Dermata Investigational Site, Saint Joseph, Missouri
  - Dermata Investigational Site, Henderson, Nevada
  - Dermata Investigational Site, Albuquerque, New Mexico
  - Dermata Investigational Site, High Point, North Carolina
  - Dermata Investigational Site, Tennessee City, Tennessee
  - Dermata Investigational Site, Austin, Texas
  - Dermata Investigational Site, College Station, Texas
  - Dermata Investigational Site, Katy, Texas

IPD SHARING:
Plan to Share IPD: No